CLINICAL TRIAL: NCT05933304
Title: Real-World Study of the Effectiveness of Moderna COVID-19 Vaccine
Brief Title: A Study of the Effectiveness of Moderna COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P901
Record Dates: First submitted 2023-07-05; First posted 2023-07-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Vaccinated Cohort: Participants who receive Moderna COVID-19 vaccine during a pre-specified time frame and meet eligibility criteria will be included in this cohort. Participants will be followed up through Electronic Health Record (EHR) for occurrence of COVID-19 outcomes until the end of the study period, or censoring events (termination of KPSC membership allowing for a 31-day gap, death, receipt of a COVID-19 vaccine).
- Unexposed Cohort: Participants in this cohort include:
  * Participants who had not received any bivalent dose but had received at least 2 doses of monovalent mRNA COVID-19 vaccine by the index date
  * Participants who never received any COVID-19 vaccine dose by the index date
  Participants will be followed up through EHR for occurrence of COVID-19 outcomes until the end of the study period, or censoring events (termination of KPSC membership allowing for a 31-day gap, death, receipt of a COVID-19 vaccine).

SUMMARY:
This is an observational cohort study to evaluate real-world vaccine effectiveness and durability of Moderna COVID-19 vaccine among a diverse population at Kaiser Permanente Southern California (KPSC).

The primary objective of this study is to evaluate the vaccine effectiveness (VE) of receipt of Moderna COVID-19 vaccine in preventing SARS-CoV-2 infection and severe COVID-19 disease.

SARS-CoV-2 infection will be defined as a positive antigen test result as well as a positive molecular diagnostic test among symptomatic or asymptomatic participants or a COVID-19 diagnosis code. Severe COVID-19 disease will be defined as COVID-19 hospitalization or mortality.

DETAILED DESCRIPTION:
This study utilized electronic healthcare data collected within the Kaiser Permanente Southern California (KPSC) integrated healthcare system which provides care to over 4.6 million individuals. Participants in this study received vaccination and were assessed for study outcomes as part of routine care. Vaccination information and study outcome status was assessed using procedure, diagnostic, and laboratory code information. Medical chart review was conducted to assess the association of severe outcomes (hospitalization and death) with COVID-19 illness.

Analyses assessing absolute vaccine effectiveness will identify participants who receive Moderna COVID vaccine from the KPSC electronic healthcare database and match them to unvaccinated participants based on age, sex, race/ethnicity, and data of vaccination (index date). Vaccinated and unvaccinated participants will then be followed-up in the database for the occurrence of study outcomes. Cox proportional hazards regression will be used to compare the relative risk of study outcomes by vaccination status.

Analyses of relative vaccine effectiveness will identify participants who receive specific dose number and formulation of Moderna COVID vaccine (Group N) from the KPSC electronic healthcare database and match them to a group of vaccinated participants with a different dose/formulation type (i.e. Group n-1). Similar matching criteria will be applied. Both groups will be followed for study outcomes and cox proportional hazards regression will be used to compare the relative risk of study outcomes by vaccination status.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at index date (participants aged 6 months through 17 years will also be included after Food and Drug Administration [FDA] authorization to vaccinate younger age groups)
* KPSC member for ≥12 months prior to index date through 14 days after the index date (allowing a 31-day gap)

Exclusion Criteria:

* Receipt of a COVID-19 vaccine other than Moderna COVID-19 vaccine prior to or on the index date
* Receipt of 2 doses of Moderna COVID-19 vaccine <24 days apart for 2-dose exposed cohort
* Receipt of any COVID-19 vaccine <14 days after the index date
* No health care utilization and no vaccination from the 2 years prior to the index date through the index date
* Occurrence of a COVID-19 outcome <14 days after the index date

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants vaccinated with Moderna COVID-19 vaccine and unvaccinated participants are included in this study.
Sampling Method: Probability Sample
Enrollment: 927004 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants With SARS-CoV-2 Infection | Up to 3 years
  SARS-CoV-2 infection is defined as a positive antigen test result as well as a positive molecular test or a COVID-19 diagnosis code.
Number of Participants With Severe COVID-19 Disease | Up to 3 years
  Severe COVID-19 disease includes COVID-19 hospitalization (hospitalization with a SARS-CoV-2 positive test or a COVID-19 diagnosis, or a hospitalization occurring ≤7 days after a SARS-CoV-2 positive test, with chart review to confirm severe COVID-19 symptoms) and COVID-19 mortality (death during COVID-19 hospitalization).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States